CLINICAL TRIAL: NCT03609398
Title: A Phase 2 Open Label Safety and Immunogenicity Study of Rift Valley Fever Vaccine, Inactivated, Dried, TSI-GSD 200, Lot 7, Run 2, in Adult Subjects at Risk of Exposure to Rift Valley Fever Virus
Brief Title: Phase 2 Safety and Immunogenicity Study of Rift Valley Fever Vaccine
Acronym: RVF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-16-12
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Rift Valley Fever
MeSH Terms: conditions — Rift Valley Fever

STUDY DESIGN:
Intervention Model Description: vaccine to be administered in 1.0mL doses SQ in the upper outer aspect of the arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RVF Vaccine (Experimental): 1.0 mL dose given SQ in upper arm
  Interventions: Biological: RVF Vaccine

INTERVENTIONS:
Biological: RVF Vaccine — 1.0 mL dose given SQ in upper arm

SUMMARY:
This study is to collect safety and immunogenicity data for an Rift Valley Fever (RVF) vaccine

DETAILED DESCRIPTION:
This study is being conducted to collect safety and immunogenicity data for the RVF vaccine, TSI-GSD 200, Lot 7, Run 2. Enrollment in this protocol is offered for personnel who enter areas where this virus is used in research or is endemic (an area where this disease process is found to occur frequently). Subjects who respond with a titer of >1:40 may participate for study duration. Rift Valley Fever Vaccine, Inactivated, Dried (TSI GSD 200) will be administered in 1.0-mL doses SQ in the upper outer aspect of the arm.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 65 years old at time of consent.
* Have RVF plaque reduction neutralization 80% titers (PRNT80) <1:10 for primary series.
* Have RVF PRNT80 (plaque reduction neutralization 80% titer) <1:40 for booster series.
* If female of childbearing potential, must agree to have a urine pregnancy test on the same day before each vaccine administration. (Exception: documented hysterectomy or ≥3 years of menopause.) The results must be negative. Females must agree not to become pregnant for 3 months after receipt of the last study treatment (vaccination).
* Be considered at risk for exposure to RVF virus and who have submitted a Request for IND Vaccines for the RVF vaccine.
* Sign and date the approved informed consent document and HIPAA Authorization.
* Have in their charts:
* medical history (including concomitant medications) within 60 days of planned first administration of vaccine
* physical examination and laboratory tests within 1 year
* previous chest radiograph results and electrocardiogram
* Be medically cleared for participation by an investigator. (Examinations and/or tests may be repeated at the discretion of the PI.)
* Be willing to return for all follow-up visits.
* Agree to report any adverse events (AEs) that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study.
* Agree to defer blood donation for 1 year after receipt of the vaccine

Exclusion Criteria:

* Have completed previous RVF vaccine study as a nonresponder (PRNT80 <1:40).
* Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the PI).
* Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
* Have confirmed HIV infection.
* Have positive pregnancy test or be breastfeeding female.
* Have any known allergies to components of the vaccine:
* Fetal rhesus monkey lung cells
* Formaldehyde
* Neomycin sulfate
* Streptomycin
* Sodium bisulfite
* Human serum albumin (HAS)
* RVF virus (Entebbe strain)
* Have administration of another vaccine or investigational product within 28 days of RVF vaccination.
* Have any unresolved AE resulting from a previous immunization.
* Have a medical condition that, in the judgment of the PI, would impact subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Local and Systemic Adverse Events and Their Relationship to the Study Vaccine | 0-28 days after each dose
  Safety assess of local and systemic adverse events and their relationship to the study vaccine. AEs will be recorded for 28 days after each dose of the vaccine for the assessment population (all subjects who receive at least one vaccination under this protocol. Subjects will be contacted by study staff via e-mail or telephone the day after vaccination (Day 1) and once per week for 4 weeks after each vaccination to discuss any reactions.
Percentage of Subjects Who Developed Titers of ≥1:40 of Per-protocol Subjects | 21-35 days after each vaccination and month 12
  Percentage of per-protocol subjects (subjects who adhered to the protocol schedule for both vaccination and blood collects) who developed titers ≥1:40 as determined by PRNT80 (plaque reduction neutralization 80% titer) after vaccination at each scheduled time point for which blood samples are drawn and over the entire study period.

SECONDARY OUTCOMES:
Frequency and Severity of Adverse Events | 0-28 days after each dose
  Frequency and severity of adverse events for the assessment population (all subjects who receive at least one vaccination under this protocol). Subjects will be contacted by study staff via e-mail or telephone the day after vaccination (Day 1) and once per week for 4 weeks after each vaccination to discuss any reactions.
Geometric Mean PRNT80 (plaque reduction neutralization 80% titer) of Per-protocol Subjects | 21-35 days after each vaccination and month 12
  Geometric mean PRNT80 (plaque reduction neutralization 80% titer) of per-protocol subjects at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.

OTHER OUTCOMES:
Geometric Mean PRNT50 (plaque reduction neutralization 50% titer) of Per-protocol Subjects | 21-35 days after each vaccination and month 12
  Geometric mean PRNT50 (plaque reduction neutralization 50% titer) of per-protocol subjects at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Special Immunization Program, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No